CLINICAL TRIAL: NCT06400901
Title: Electrophysiology Based Brain Network Study on Deep Brain Nuclei LFP and Cortical EEG During the Recovery From General Anesthesia
Brief Title: Analysis of Deep Brain Nuclei LFP and Cortical EEG Signals During the Recovery From General Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Xin Ma, MD, Attending Anesthesiologist, Ruijin Hospital
Other Study IDs: 2023(426)
Record Dates: First submitted 2024-04-16; First posted 2024-05-06 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Deep Brain Stimulation Surgery; Electrophysiology; General Anesthesia; Consciousness, Loss of
Keywords: cortex EEG; deep brain nuclei; local field potentiation; propofol
MeSH Terms: conditions — Unconsciousness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No interventions — No interventions were given to patients except for the deep brain stimulation surgery they originally planned to take

SUMMARY:
The correlations of deep brain nuclei firing and cerebral cortex activity during recovery from general anesthesia is unclear. In this study, the local field potential (LFP) from the deep brain nuclei and the scalp electroencephalogram (EEG) of the frontal cortex were recorded from patients undergoing deep brain stimulation (DBS) surgery during the recovery from general anesthesia, in order to explore the changes and relevance of deep brain nuclei firing and cortex activity during the recovery of consciousness from general anesthesia .

DETAILED DESCRIPTION:
The recovery of consciousness during the emergence from general anesthesia is an important part of general anesthesia. Previous studies have found that the recovery of consciousness is not a passive process of drug metabolism, but involves the activation of functional neural networks in the brain. However, the temporal-spatial dynamics of different brain regions, including deep brain nuclei and the cortex, during recovery from general anesthesia have not been elucidated.

At present, thanks to the perceptible function of the new generation of deep brain stimulation (DBS) equipment, the local field potential (LFP) of deep brain nuclei can be recorded in real time during the patient's recovery from general anesthesia after DBS surgery. This study will simultaneously record the electrophysiological signals of the patient's deep brain nuclei LFP and cortical EEG signals, and analyze the differences and correlations between the deep brain nuclei LFP and the cortical EEG characteristics during recovery from general anesthesia. This provides evidence for understanding how subcortical deep brain nuclei are involved in the recovery of general anesthesia, and provides clues for solving the mystery of consciousness.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* ASA (American Society of Anesthesiologists) classification I-III
* Those who meet the indications for DBS surgery
* Right-handed with normal listening and speaking abilities
* The patient signs the informed consent form and cooperates with the researchers

Exclusion Criteria:

* Patients with cognitive impairment [Montreal Cognitive Assessment (MoCA) score less than 26 points];
* Patients with severe depression [Beck Depression Inventory (BDI-II) score greater than or equal to 25 points];
* Patients with important organs dysfunction, such as heart, lungs, liver, and kidneys; or patients with unstable vital signs;
* Patients who are expected to enter the ICU after surgery;
* Patients who are alcoholic, alcohol dependent or drug dependent;
* Patients who have received general anesthesia one month before surgery, patients who are known to be allergic to general anesthetics;
* The DBS surgery exceeds 4 hours;
* Patients who are pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the surgical indications and voluntarily undergo DBS surgery at the Functional Neurosurgery Department of Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine from April 2024 until October 2026.
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Changes in the Local Field Potential from the Deep Brain Nuclei and the Scalp Electroencephalogram of the Frontal Cortex. | 2 hours.
  Number of participants with changes in the local field potential from the deep brain nuclei and the scalp electroencephalogram of the frontal cortex during recovery of consciousness from general anesthesia. The recovery of consciousness is defined as the patient can follow the experimenter's verbal command to open mouth and extubate the endotracheal tube.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang Y, Hu K, Green AL, Ma X, Gillies MJ, Wang S, Fitzgerald JJ, Pan Y, Martin S, Huang P, Zhan S, Li D, Tan H, Aziz TZ, Sun B. Dynamic changes in rhythmic and arrhythmic neural signatures in the subthalamic nucleus induced by anaesthesia and tracheal intubation. Br J Anaesth. 2020 Jul;125(1):67-76. doi: 10.1016/j.bja.2020.03.014. Epub 2020 Apr 24. PMID 32336475
- [Result] Huang Z, Vlisides PE, Tarnal VC, Janke EL, Keefe KM, Collins MM, McKinney AM, Picton P, Harris RE, Mashour GA, Hudetz AG. Brain imaging reveals covert consciousness during behavioral unresponsiveness induced by propofol. Sci Rep. 2018 Sep 4;8(1):13195. doi: 10.1038/s41598-018-31436-z. PMID 30181567